CLINICAL TRIAL: NCT02046226
Title: A Prospective, Randomized, Single-center Pilot Study of the OxyGenesys™ Dissolved Oxygen Dressing to Improve Chronic Wound Healing After Revascularization for Critical Limb Ischemia
Brief Title: Dissolved Oxygen Dressing to Improve Chronic Wound Healing After Revascularization for Critical Limb Ischemia
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: inability to meet enrollment goals in this subject population
Sponsor: Halyard Health (Industry)
Collaborators: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 100-13-0001
Record Dates: First submitted 2014-01-23; First posted 2014-01-27 (Estimated); Results first posted 2015-10-12 (Estimated); Last update posted 2015-10-12 (Estimated); Status verified 2014-11

CONDITIONS: Critical Limb Ischemia
Keywords: Critical Limb Ischemia; Non Healing Wounds; Diabetic Wounds; Foot Ulcers
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia; Foot Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- OxyGenesys(TM) Dissolved Oxygen Dressing (Experimental): OxyGenesys(TM) Dissolved Oxygen Dressing
  Interventions: Device: Oxygenesys(TM) Dissolved Oxygen Dressing
- Standard Wound Care (No Intervention): Standard wound care using gauze dressings per institutional standard of care.

INTERVENTIONS:
Device: Oxygenesys(TM) Dissolved Oxygen Dressing — OxyGenesys(TM) Dissolved Oxygen Dressing
  Arms: OxyGenesys(TM) Dissolved Oxygen Dressing

SUMMARY:
A Prospective, Randomized, Single-center Pilot Study of The OxyGenesys(TM) Dissolved Oxygen Dressing to Improve Chronic Wound Healing after REvascularization for Critical Limb Ischemia.

DETAILED DESCRIPTION:
A Prospective, Randomized, controlled pilot study enrolling up to 50 subjects at a singe investigational site in the US. Subjects with atherosclerotic peripheral arteria disease (PAD) presenting with critical limb ischemia (CLI) and one or more non-healing lower extremity arterial insufficiency ulcers who are suitable candidates for revascularization procedures (endovascular or surgical) will be randomized 1:1 to:

* Wound care with the use of OxyGenesys(TM) Dissolved Oxygen Dressing, or
* Standard Wound Care procedures

An initial study phase will enroll up to 20 subjects (10 in each arm). Pending results of the initial study phase, the study may continue to enroll until up to 50 subjects (25 in each arm) have been enrolled.

All subjects will be followed clinically and receive wound evaluation at 1, 3, and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant female >=21 years of age
* A clinical diagnosis of critical limb ischemia (CLI) with Rutherford classification stage 5
* One or more chronic ulcers with a presumed etiology of arterial insufficiency and duration >2 weeks. The target ulcer is defined as the highest-grade ulcer (Wagner's classification) at initial evaluation. For wounds with identical grading, the largest wound is the index wound
* The patient or legally authorized representative is willing to provide informed consent and comply with specified follow-up evaluations
* Undergoing intervention for infrainguinal or infrapopliteal artery disease (below the femoral artery bifurcation and above the ankle joint)
* The index procedure resulted in successful revascularization. For endovascular procedures, successful revascularization is defined as complete revascularization of the target ulcer culprit vessels according to the angiosome treatment strategy, with a final percent diameter stenosis >50% and improved distal flow by angiography following the procedure. For surgical procedures, successful revascularization is defined as a patent graft and improved distal flow following the procedure.

Exclusion Criteria:

* Pregnant or nursing patients and those who plan pregnancy in the period up to 1 year following index procedure. Female patients of child-bearing potential must have a negative pregnancy test done within 7 days prior to index procedure.
* Rutherford classification stage 0,1,2,3,4, or 6
* Target wound duration <2 weeks
* Presence of frank gangrene (Wagner classification grade 4 or 5), major tissue loss (severe/extensive necrosis), or unsalvageable limb (extensive ischemic ulceration beyond the transmetatarsal level anticipated to require major amputation after the index procedure)
* Previous or planned surgical or interventional procedure within 6 months before or 30 days after the index procedure, or any previous or planned target limb amputation.
* Active local or systemic infection
* Patients with ulcers judged by the examining physician to have a primary etiology other than ischemic arterial disease (e.g., venous related, decubitus, or other [goug, pyoderma gangrenosum, necrobiosis lipoidica, vitamin B12 deficiency])
* Renal failure or chronic kidney disease with estimated glomerular filtration rate (eGFR <30 ml/min/1.7sm sq. within 30 days of the index procedure or treated with dialysis)
* Severly decreased cardiac output
* Uncontrolled hyperglycemia
* Patients with a known other medical illness or known history of substance abuse that may cause non-compliance with the protocol, confound data interpretation, or is associated with a life expectancy of less than 1 year
* Patient is currently participating (or has participated in the last 30 days) in a study of any other investigational treatment.
* Ulcer treatment with normothermic or hyperbaric oxygen therapy, recombinant or autologous growth factor products, or use of enzymatic debridement
* Concomitant medications such as corticosteroids, immunosuppressive medications, or chemotherapy
* Acute thrombus in the target limb

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2013-08; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Mena-Hurtado, MD, Principal Investigator — Yale University; David T Curd, MS, Study Director — Kimberly-Clark Corporation
Locations (1):
- Yale New Haven Hospital, New Haven, Connecticut, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The randomization of subjects to either of the two treatments (OxyGenesys(TM) Dissolved Oxygen Dressing or standard wound care using gauze dressings per institutional standard of care) in this study was not indicated on each of the case report forms of the seven subjects enrolled.
Groups:
- All Study Participants: The seven study subjects were treated with OxyGenesys(TM) Dissolved Oxygen Dressing or standard wound care using gauze dressings per institutional standard of care. The randomization of these subjects to either of these treatments was not indicated in each of the case report forms.
Period: Overall Study
Arm/Group | All Study Participants
Started | 7
Completed | 0
Not Completed | 7
Not completed — Lost to Follow-up | 7

BASELINE CHARACTERISTICS:
Arm/Group | All Study Participants
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants] — Not applicable - subjects' ages were not collected.
  Participants
    <=18 years | NA — Study subjects' ages were not collected.
    Between 18 and 65 years | NA — Study subjects' ages were not collected.
    >=65 years | NA — Study subjects' ages were not collected.
Sex: Female, Male [Count of Participants; unit: Participants] — Not applicable - subjects' gender information was not recorded.
  Participants
    Female | NA — Study subjects' gender information was not recorded.
    Male | NA — Study subjects' gender information was not recorded.

OUTCOME MEASURES:

1. Primary Outcome: Rate of Wound Healing
Description: Percentage reduction in target wound area (length x width).
Time Frame: 3 months
Population: Study subjects were not available to provide data when the primary outcome was to be reported, and thus there are no primary outcome data to report.
Arm/Group | OxyGenesys(TM) Dissolved Oxygen Dressing | Standard Wound Care
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Incidence of Complete Wound Closure
Description: number of wounds undergoing complete reepithelialization without drainage or dressing requirements, maintained for at least 2 weeks.
Time Frame: 3 months
Population: Study subjects were not available to provide data when the secondary outcome was to be reported, and thus there are no secondary outcome data to report.
Arm/Group | OxyGenesys(TM) Dissolved Oxygen Dressing | Standard Wound Care
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: Adverse events were not collected/assessed for the study subjects.
Groups:
- All Study Participants: The seven study subjects were treated with OxyGenesys(TM) Dissolved Oxygen Dressing or standard wound care using gauze dressings per institutional standard of care. The randomization of these subjects to either of these treatments was not indicated on each case report form.
Arm/Group | All Study Participants
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
An agreement between Sponsor and Investigator(s) in the final form of abstracts and articles shall be obtained within an appropriate time frame of 60 days. Any and all information supplied or obtained during this study by or on behalf of any party involved in the study (in whatever form) shall be treated as confidential, shall not be disclosed to any third party unless with the prior written consent of the Sponsor in each case.